CLINICAL TRIAL: NCT03912155
Title: Multi-scale Analysis of Physiological and Pathological Brain Networks by Simultaneous EEG-MEG-SEEG Recordings
Brief Title: Multi-scale Analysis of Physiological Brain Networks
Acronym: SCALES
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-51; 2018-A02363-52 RCB (Registry Identifier: APHM)
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
Keywords: MEG; EEG; SEEG
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 20 patients per presumed location of the epileptogenic zone (see experimental plan) for a total of 120 patients, including 30 minors. For patients, a MEG-EEG-SEEG examination during the SEEG exploration period.
  Interventions: Other: Multi-scale analysis of physiological brain networks
- Controles: For the control population, 120 control subjects, including 30 minors, that is to say as many as patients. For control subjects, a MEG-EEG exam.
  Interventions: Other: Multi-scale analysis of physiological brain networks

INTERVENTIONS:
Other: Multi-scale analysis of physiological brain networks — It will be simultaneously record the surface EEG, the MEG and in patients only the intracerebral EEG (SEEG). In the case of SEEG with micro contacts, these additional signals will also be recorded in parallel and will provide greater sensitivity to high frequency activities. The physiological networks will be studied in patients thanks to stimulations (external or intracerebral) carried out within the framework of the functional cartography, and the pathological networks thanks to measures in state of rest. For external stimulation protocols, it will be constitute a reference base in MEG and EEG alone (non-invasive) on control subjects.

SUMMARY:
The SEEG implantation is performed on purely clinical criteria for preoperative diagnosis. Magnetoencephalography and EEG are purely passive techniques that do not involve any additional risk. This project is a continuation of an existing project in which it was demonstrated the feasibility of simultaneous SEEG and MEG/EEG recordings.

DETAILED DESCRIPTION:
Brain function is based on the communication between sets of neurons at different spatial and temporal scales. The dysfunction of these networks is thus at the origin of several brain pathologies, including epilepsy. The recent improvement in recording methods paves the way for better characterization of brain networks, with several spatial and temporal resolutions, depending on the techniques used.

Still, several key points remain outstanding. First, several mechanisms can underlie the interaction between brain regions, and it remains to determine the most relevant tools in practice to quantify them. Second, there are difficulties in extracting these networks from surface recordings. The best strategies for studying these interactions in a non-invasive way therefore remain to be defined.

It will be propose to answer these questions based on simultaneous surface (magneto-encephalography/ electroencephalography) and depth (intracerebral stereotactic EEG, SEEG) recordings, a technique it was developed by the team of Marseille, in patients undergoing preoperative epilepsy assessment.

The primary objective is to find, among all the mechanisms of interaction between brain regions, which are most relevant in describing physiological and pathological brain networks.

The secondary objective is to test whether the visible coupling information at depth can be found from surface data (EEG, MEG) only. To do this, it will be compare the surface results with the SEEG results.

The SEEG implantation is performed on purely clinical criteria for preoperative diagnosis. Magnetoencephalography and EEG are purely passive techniques that do not involve any additional risk. This project is a continuation of an existing project in which we have demonstrated the feasibility of simultaneous SEEG and MEG/EEG recordings.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients

  * Patients for whom intracerebral electrode implantation is in progress as part of the pre-surgical evaluation of their drug-resistant partial epilepsy.
  * Patient informed, expressing his non-opposition (or legal representative (s), affiliated to a social security scheme
  * The medical examination is carried out as part of the medical follow-up of these patients
* Inclusion criteria for control subjects

  • Informed subject, expressing his non-opposition or legal representative, affiliated to a social security scheme
* Exclusion Criteria:

Minors under 12 years

* Pregnant or lactating women,
* The adults under guardianship or under the protection of justice
* Non-beneficiaries of a social security scheme
* Persons deprived of their liberty by a judicial or administrative decision
* Absence of informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients will be recruited in the Service of Epileptology and Cerebral Rhythmology of the Timone. Only major and minor control subjects will be recruited following the announcement of the experience by posting on different sites or other appropriate means of communication.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Rate of epileptic discharges | 2 hours
  Measurement of epileptic activity by electroencephalogram
Rate of epileptic discharges | 2 hours
  Measurement of epileptic activity by magneto-encephalography
Rate of epileptic discharges | 2 hours
  Measurement of epileptic activity by intracerebral stereotactic electroencephalogram

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France